CLINICAL TRIAL: NCT03027492
Title: Gynaecological Disorders in Patients With Not-celiac Wheat Sensitivity
Brief Title: Gynaecological Disorders in Not-celiac Wheat Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Pasquale Mansueto, MD, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ACPM15
Record Dates: First submitted 2016-12-30; First posted 2017-01-23 (Estimated); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Non-celiac Wheat Sensitivity
Keywords: Non-celiac Wheat Sensitivity; gynaecological disorders; gluten-free diet
MeSH Terms: interventions — Diet, Gluten-Free

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1. NCWS retrospective patients (Active Comparator): The clinical charts of NCWS female patients attending the outpatient centers of the Department of Internal Medicine at the University Hospital of Palermo and the Department of Internal Medicine of the Hospital of Sciacca will be reviewed with a retrospective method. They had all been diagnosed with NCWS between January 2001 and June 2011 and included in a previously published study. These charts included specific sections for associated gynaecological disorders. Incomplete clinical charts will be excluded. All the patients will be evaluated at baseline (i.e. at diagnosis) and after at least a 6-months period of gluten-free diet.
  Interventions: Other: Gluten free diet
- 2. CD retrospective control patients (Active Comparator): To compare the presence and characteristics of gynaecological disorders in NCWS female patients, a control group of CD female patients had been randomly chosen by a computer-generated method from female patients diagnosed during the same period (2001-2011) and age- (+2 years) matched with the NCWS female patients. Similar to NCWS patients, also this control group was asked for gynaecological disorders and the answers reported in the patients clinical charts. All the patients will be evaluated at baseline (i.e. at diagnosis) and after at least a 6-months period of gluten-free diet.
  Interventions: Other: Gluten free diet
- 3. IBS retrospective control patients (Active Comparator): To compare the presence and characteristics of gynaecological disorders in NCWS female patients, a control group of IBS female patients had been randomly chosen by a computer-generated method from female subjects diagnosed during the same period (2001-2011) and age- (+2 years) matched with the NCWS female patients. Similar to NCWS patients, also this control group was asked for gynaecological disorders and the answers reported in the patients clinical charts. All the patients will be evaluated at baseline (i.e. at diagnosis) and after at least a 6-months period of gluten-free diet.
  Interventions: Other: Gluten free diet
- 4. NCWS prospective patients (Active Comparator): The investigators prospectively will survey adult female patients with functional gastroenterological symptoms according to the Rome III criteria, and a suspected diagnosis of NCWS. The patients will be recruited between January 2017 and January 2018 at the same 2 centers. Most of the patients will be referred owing to gastrointestinal and extraintestinal symptoms, the onset of which, they reported, could be related to wheat ingestion. In addition, patients will be asked about the presence and characteristics of gynaecological disorders using an ad hoc questionnaire. All the patients will be evaluated at baseline (i.e. at diagnosis) and after at least a 6-months period of gluten-free diet.
  Interventions: Other: Gluten free diet
- 5. CD prospective control patients (Active Comparator): To compare the presence and characteristics of gynaecological disorders in NCWS female patients, a control group of CD female patients will be randomly chosen by a computer-generated method from female subjects diagnosed during the same period (2017-2018) and age- (+2 years) matched with the NCWS female patients. Similar to NCWS patients, also this control group will be asked for gynaecological disorders and the answers reported in the patients clinical charts. All the patients will be evaluated at baseline (i.e. at diagnosis) and after at least a 6-months period of gluten-free diet.
  Interventions: Other: Gluten free diet
- 6. IBS prospective control patients (Active Comparator): To compare the presence and characteristics of gynaecological disorders in NCWS female patients, a control group of IBS female patients will be randomly chosen by a computer-generated method from female subjects diagnosed during the same period (2017-2018) and age- (+2 years) matched with the NCWS female patients. Similar to NCWS patients, also this control group will be asked for gynaecological disorders and the answers reported in the patients clinical charts. All the patients will be evaluated at baseline (i.e. at diagnosis) and after at least a 6-months period of gluten-free diet.
  Interventions: Other: Gluten free diet

INTERVENTIONS:
Other: Gluten free diet — The investigators will evaluate the modification of gynaecological disorder after a gluten (wheat)-free diet.

SUMMARY:
In the last few years, a new clinical entity has emerged which includes patients who consider themselves to be suffering from problems caused by wheat and/or gluten ingestion, even though they do not have celiac disease (CD) or wheat allergy. This clinical condition has been named non-celiac gluten sensitivity (NCGS), although in a recent article, the investigators suggested the term "non-celiac wheat sensitivity" (NCWS), because it is not known to date what component of wheat actually causes the symptoms. The clinical picture of NCWS is characterized by combined gastrointestinal (bloating, abdominal pain, diarrhea and/or constipation, nausea, epigastric pain, gastroesophageal reflux, aphthous stomatitis) and very different extra-intestinal and systemic manifestations (headache, depression, anxiety, 'foggy mind,' tiredness, dermatitis or skin rash, fibromyalgia-like joint/muscle pain, leg or arm numbness, and anemia). Nowadays, there no data about a possible relationship between gynaecological disorders and food ingestion and food allergy/intolerance. Therefore, the aims of the present study are to investigate 1) the prevalence and characteristics of gynaecological disorders in NCWS patients compared to CD and irritable bowel syndrome (IBS) controls, and 2) the modification of such disorders in NCWS patients after a gluten (wheat)-free diet.

DETAILED DESCRIPTION:
In the last few years, a new clinical entity has emerged which includes patients who consider themselves to be suffering from problems caused by wheat and/or gluten ingestion, even though they do not have CD or wheat allergy. This clinical condition has been named non-celiac gluten sensitivity (NCGS), although in a recent article, the investigators suggested the term "non-celiac wheat sensitivity" (NCWS), because it is not known to date what component of wheat actually causes the symptoms. Other areas of doubt in NCWS regard its pathogenesis, while some papers reported intestinal immunologic activation, others linked NCWS to the dietary short chain carbohydrate (fermentable oligo-di-monosaccharides and polyols, FODMAPs) load. The investigators recently demonstrated that higher proportions of patients with NCWS develop autoimmune disorders, are antinuclear antibodies (ANA) positive, and show DQ2/DQ8 haplotypes compared with patients with IBS, supporting an immunologic involvement in NCWS. The clinical picture of NCWS is characterized by combined gastrointestinal (bloating, abdominal pain, diarrhea and/or constipation, nausea, epigastric pain, gastroesophageal reflux, aphthous stomatitis) and very different extra-intestinal and systemic manifestations (headache, depression, anxiety, 'foggy mind,' tiredness, dermatitis or skin rash, fibromyalgia-like joint/muscle pain, leg or arm numbness, and anemia). Nowadays, there no data about a possible relationship between gynaecological disorders (i.e. menstrual cycle alterations, vaginitis, recurrent vulvovaginitis, recurrent cystitis, chronic pelvic pain, recurrent pregnancy loss, infertility) and food ingestion and food allergy/intolerance. Therefore, the aims of the present study are to investigate 1) the prevalence and characteristics of gynaecological disorders in NCWS patients compared to CD and IBS controls, and 2) the modification of such disorders in NCWS patients after a gluten (wheat)-free diet.

ELIGIBILITY:
Inclusion Criteria:

To diagnose NCWS the recently proposed criteria will be adopted. All the patients will meet the following criteria:

* negative serum anti-transglutaminase (anti-tTG) and anti-endomysium (EmA) immunoglobulin (Ig)A and IgG antibodies
* absence of intestinal villous atrophy
* negative IgE-mediated immune-allergy tests to wheat (skin prick tests and/or serum specific IgE detection)
* resolution of the IBS symptoms on standard elimination diet, excluding wheat, cow's milk, egg, tomato, chocolate, and other self-reported food(s) causing symptoms
* symptom reappearance on double-blind placebo-controlled (DBPC) wheat challenge. As the investigators previously described in other studies, DBPC cow's milk protein challenge and other "open" food challenges will be performed too.

To diagnose CD the standard criteria will be adopted. All the patients will meet the following criteria:

* positive serum anti-transglutaminase (anti-tTG) and anti-endomysium (EmA) immunoglobulin (Ig)A and IgG antibodies
* presence of intestinal villous atrophy.

To diagnose IBS the standard Rome II (for retrospective patients) and Rome III (for prospective patients) Criteria will be adopted. None of these subjects improved on an elimination diet without wheat, cow's milk, egg, tomato, or chocolate.

Exclusion Criteria:

For NCWS diagnosis it will be evaluated the following exclusion criteria:

* positive EmA in the culture medium of the duodenal biopsies, also in the case of normal villi/crypts ratio in the duodenal mucosa
* self-exclusion of wheat from the diet and refusal to reintroduce it before entering the study
* other previously diagnosed gastrointestinal disorders
* other previously diagnosed gynaecological disorders
* nervous system disease and/or major psychiatric disorder
* physical impairment limiting physical activity.

Ages: 15 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2001-01-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Gynaecological disorders in NCWS female patients at baseline | Up to 200 months
  Prevalence of gynaecological disorders in retrospective and prospective NCWS female patients, compared to retrospective and prospective CD and IBS female patients.

SECONDARY OUTCOMES:
Gynaecological disorders in NCWS female patients after gluten-free diet. | Change from baseline at 6 months of gluten-free diet
  Gynaecological disorders evaluation after at least 6 months of gluten-free diet after the NCWS diagnosis, by visual analogic scales, specific questionnaire, and clinical examination, both in retrospective and prospective NCWS female patients.
Pap smear in NCWS female patients after gluten-free diet. | Change from baseline at 6 months of gluten-free diet
  PAP smear after at least 6 months of gluten-free diet after the NCWS diagnosis, both in retrospective and prospective NCWS female patients.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Carroccio, PhD, Study Director — University of Palermo
Locations (2):
- Italy (2):
  - Department of Internal Medicine, Giovanni Paolo II Hospital of Sciacca, Sciacca, Agrigento
  - Department of Internal Medicine, University Hospital of Palermo, Palermo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Di Liberto D, Mansueto P, D'Alcamo A, Lo Pizzo M, Lo Presti E, Geraci G, Fayer F, Guggino G, Iacono G, Dieli F, Carroccio A. Predominance of Type 1 Innate Lymphoid Cells in the Rectal Mucosa of Patients With Non-Celiac Wheat Sensitivity: Reversal After a Wheat-Free Diet. Clin Transl Gastroenterol. 2016 Jul 7;7(7):e178. doi: 10.1038/ctg.2016.35. PMID 27388423
- [Result] Mansueto P, D'Alcamo A, Seidita A, Carroccio A. Food allergy in irritable bowel syndrome: The case of non-celiac wheat sensitivity. World J Gastroenterol. 2015 Jun 21;21(23):7089-109. doi: 10.3748/wjg.v21.i23.7089. PMID 26109796
- [Result] Carroccio A, Soresi M, D'Alcamo A, Sciume C, Iacono G, Geraci G, Brusca I, Seidita A, Adragna F, Carta M, Mansueto P. Risk of low bone mineral density and low body mass index in patients with non-celiac wheat-sensitivity: a prospective observation study. BMC Med. 2014 Nov 28;12:230. doi: 10.1186/s12916-014-0230-2. PMID 25430806
- [Result] Mansueto P, Seidita A, D'Alcamo A, Carroccio A. Non-celiac gluten sensitivity: literature review. J Am Coll Nutr. 2014;33(1):39-54. doi: 10.1080/07315724.2014.869996. PMID 24533607
- [Result] Carroccio A, Rini G, Mansueto P. Non-celiac wheat sensitivity is a more appropriate label than non-celiac gluten sensitivity. Gastroenterology. 2014 Jan;146(1):320-1. doi: 10.1053/j.gastro.2013.08.061. Epub 2013 Nov 22. No abstract available. PMID 24275240
- [Result] Carroccio A, Mansueto P, D'Alcamo A, Iacono G. Non-celiac wheat sensitivity as an allergic condition: personal experience and narrative review. Am J Gastroenterol. 2013 Dec;108(12):1845-52; quiz 1853. doi: 10.1038/ajg.2013.353. Epub 2013 Nov 5. PMID 24169272
- [Result] Carroccio A, Mansueto P, Iacono G, Soresi M, D'Alcamo A, Cavataio F, Brusca I, Florena AM, Ambrosiano G, Seidita A, Pirrone G, Rini GB. Non-celiac wheat sensitivity diagnosed by double-blind placebo-controlled challenge: exploring a new clinical entity. Am J Gastroenterol. 2012 Dec;107(12):1898-906; quiz 1907. doi: 10.1038/ajg.2012.236. Epub 2012 Jul 24. PMID 22825366